CLINICAL TRIAL: NCT05537662
Title: External Sensing and Neuromodulation to Assess Diabetic Pain Outcomes
Brief Title: External Sensing and Neuromodulation to Assess Diabetic Pain Outcomes (XANADO)
Acronym: XANADO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10458
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain
Keywords: ABT-CIP-10458; Chronic Pain; Neuromodulation System; SCS; Diabetic Pain; DRG
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subjects using Neuromodulation Therapy (SCS or DRG) (Experimental): Patients will trial standard of care neuromodulation therapy (SCS or DRG), and if successful will proceed to a permanent implant.
  Interventions: Device: Standard of care neuromodulation therapy (SCS or DRG)

INTERVENTIONS:
Device: Standard of care neuromodulation therapy (SCS or DRG) — Standard SCS or DRG therapy

SUMMARY:
This is a prospective, longitudinal, single-center, non-randomized, open-label, post-market clinical feasibility study to assess the efficacy of neuromodulation therapies (SCS and DRG) for chronic pain patients with diabetes and investigate whether physical and physiological data collected from diabetic and pre-diabetic chronic pain patients is predictive of subjective patient-reported outcomes (PROs) and of adjustments in patient care. These assessments will be made prior to, during, and after the trial of the SCS or DRG system. The study will be carried out in the United States at a single site.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to any clinical investigation-related procedure.
2. Subject is at least 18 years of age or older at the time of enrollment.
3. Subject's scheduled trial duration for the Abbott neuromodulation system is at least 7 days.
4. Subject is scheduled to undergo trial of an Abbott neuromodulation system for chronic intractable back and/or leg pain at least 7 days after enrollment and commencement of the baseline data collection period.
5. Subject agrees to take an A1C screening test prior to study enrollment and has a confirmed HbA1C level ≥ 5.7%.
6. Subject has a baseline (with no stimulation) pain NRS of ≥ 6.
7. Subject is willing to cooperate with the study requirements including completion of all office visits.
8. Subject agrees to wear the wearable sensing devices (Fitbit® and Freestyle Libre).
9. Subject agrees to answer questionnaires regularly for the duration of the study.

Exclusion Criteria:

1. Subject is enrolled, or intends to participate, in a competing or confounding clinical study, as determined by Abbott.
2. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
3. Subject is part of a vulnerable population.
4. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation results.
5. Subject has a current diagnosis of a coagulation disorder, bleeding diathesis, progressive peripheral vascular disease, post-herpetic neuralgia.
6. Subject has, or is scheduled to receive, implantation of another neuromodulation system (e.g. DRG or SCS system or intrathecal pump) to address their chronic pain.
7. Subject has already participated in a SCS trial period before enrolling in the study.
8. Subject engages in a profession or other activity that could be damaging to the wearable sensors, as determined by the investigator.
9. Subject has a physical condition that makes it difficult to wear the wearable sensors, as determined by the investigator.
10. Subject has tremors (e.g. Parkinson's disease or Familial tremors).
11. Subject has sleep/wake schedule that would present a challenge in completing all clinical site visits or in use of the wearable devices and engagement in the surveys via the mobile device.
12. Subject is bedridden.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The mean change in pain scores measured by the Numerical Rating Scale (NRS) at baseline and follow up at 3 months | At 3 month
  Change in pain scores measured by the NRS at baseline and follow up study visits at 3 months.
The mean change in pain scores measured by the Numerical Rating Scale (NRS) at baseline and follow up at 6 months | At 6 month
  Change in pain scores measured by the NRS at baseline and follow up study visits at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No